CLINICAL TRIAL: NCT04860869
Title: Endocrine, Metabolic and Microbiome Influence on the Post-acute Sequelae SARS-CoV-2 (PASC)
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0361
Record Dates: First submitted 2021-03-03; First posted 2021-04-27 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Covid19
Keywords: cognitive impairment; fatigue
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- symptomatic post-acute sequelae SARS-CoV-2 (PASC): Patients with post-acute sequelae SARS-CoV-2 (PASC) after COVID-19 infection
- non-symptomatic post-COVID: Patients with that recovered without lingering symptoms after being infected with COVID

SUMMARY:
The aim of this study is characterize the endocrine, metabolic and microbiomes of patients with post-acute sequelae SARS-CoV-2 infection (PASC) and patients that have recovered from COVID without lingering symptoms.

DETAILED DESCRIPTION:
The onset of the COVID-19 pandemic has led to a subset of patients that, once recovered from the acute infection, also experience an intractable and debilitating set of lingering symptoms termed post-acute sequelae SARS-CoV-2 infection (PASC). The most common symptoms include anxiety, shortness of breath, continued loss of the sense of smell and taste, loss of appetite with subsequent weight loss, sleep difficulties, severe fatigue, cognitive dysfunction (foggy brain) and increased frailty. These patients frequently present to the emergency room looking for symptom management because they are unable to perform normal activities of daily living and maintain job performance. Thus, it is critical to characterize the baseline endocrine, metabolic, inflammatory and microbiome alterations in the post-COVID syndrome patients to better identify and manage the symptoms to prevent potential long-term health consequences.

University of Texas Medical Branch (UTMB) has established a post-COVID clinic for management of these patients, but it is recognized that a more complete clinical picture of the underlying mechanisms driving these lingering symptoms is needed.

Persistent and long-lasting health problems are common in patients after COVID-19 infection. In a recent study of patients that had been hospitalized with COVID-19, two months after discharge, 87% reported at least one lingering symptom (joint pain, fatigue, breathing issues, etc), more than 50% reported more than three lingering issues, and over 40% reported a reduction in their of quality of life. Another study found that at 1-month after hospitalization for COVID-19, 74% reported persistent issues related to shortness of breath and a decrease in both physical and mental health. Preliminary data from the UTMB Post-COVID Recovery clinic agree with these two recent reports. In a recent study, 1 1/2 months after COVID-19 diagnosis, patients reported on average 10 of the 18 common symptoms (with 90% having chest pain, 87% dyspnea, 75% fatigue, and 90% with cognitive changes). While the previous studies examined patients that had severe COVID-19 infections, >50% of the patients were never hospitalized, yet have numerous persistent symptoms. This has serious implications for the ability of patients to return to work, downstream effects on mental health due to sometimes drastic lifestyle and work capacity changes, and the ability to engage in activities or hobbies enjoyed prior to COVID-19 illness.

Notably, the cluster of symptoms associated with PASC include profound fatigue and cognitive dysfunction, which are strikingly consistent with a syndrome that the investigators clinical research team has described in patients after traumatic brain injury (TBI) designated Brain Injury Associated Fatigue and Altered Cognition (BIAFAC). Over the last 12 months the investigators have reported the characteristics of BIAFAC syndrome. In particular, TBI patients with BIAFAC present with lingering and profoundly debilitating symptoms including severe fatigue, cognitive dysfunction (foggy brain), sleep disturbances, and the inability to perform activities of daily living that persist for years post-injury. Mechanistically the investigators have explored the role of the gut microbiome discovering altered communities in TBI patients in long-term care facilities compared with controls. The investigators also established that many TBI patients with BIAFAC also present with abnormal growth hormone (GH) secretion, and when treated with recombinant GH, a majority of patients have significant improvement of both fatigue and impaired cognition. While studies are underway to understand the details of the mechanism causing BIAFAC and why GH treatment alleviates symptoms in these patients, the investigators are intrigued that the symptom phenotype with PASC patients overlaps with many BIAFAC symptoms. It is possible that PASC may be addressed through similar treatment strategies including the potential for prebiotic/probiotic enhancement of microbiome health.

In the current pilot proposal, the investigators will characterize the baseline endocrine, metabolic, inflammatory and gut microbiome alterations in PASC patients and patients who recovered without lingering symptoms from COVID infection. These patients will be compared to the investigators extensive database of BIAFAC patients and normal controls. From this critical baseline data, the investigators will develop carefully defined clinical research trials that will test potential treatments for alleviating the syndrome. The investigators hypothesize that an imbalanced endocrine axis stemming from COVID-19 infection leads to metabolic, inflammatory and microbial dysregulation resulting in the onset of persistent post-COVID symptoms.

Specific Aims

Specific Aim 1: Characterize the baseline physiological measures of endocrine function, metabolism, inflammation, and composition of the gut and nasal microbiome of patients reporting symptoms of PASC.

Specific Aim 2: Assess baseline neuropsychological measures of fatigue, sleep, and cognition for patients reporting symptoms of PASC.

Specific Aim 3: Correlate physiological and neuropsychological measures of PASC and compare those measures to the investigators extensive database of BIAFAC patients and normal controls.

Specific Aim 4: Characterize the microbiome of patients with PASC and compare to: a)our database of healthy control subjects, b) our database of symptomatic BIAFAC patients, c) new collected samples of patients with a history of COVID who did not develop PASC.

ELIGIBILITY:
COVID Non-Symptomatic controls (nPASC)

Inclusion criteria

1. Male or female with a history of COVID with diagnosis confirmed by PCR test.
2. Minimum of 6 months since diagnosis of COVID by PCR test.
3. Ages 18 to 80 years.
4. Participant is willing and able to give informed consent for participation in the study.

Exclusion criteria

1. Current COVID infection.
2. Unable to walk unassisted.
3. Significant heart, liver, kidney, blood or respiratory disease as determined by Principal Investigator.
4. Uncontrolled diabetes mellitus.
5. Any history of a recently (12 months) diagnosed cancer other than a skin cancer (excluding melanoma).
6. Current alcohol or drug abuse.
7. History of psychosis.
8. Pregnancy or become pregnant during the trial.
9. Subjects who are being managed with narcotics will be excluded as the effects of central nervous system depressants may interfere with study test results.
10. Other medical condition or medication administration deemed exclusionary by the study investigators.

COVID Symptomatic Subjects (PASC)

Inclusion Criteria:

1. Male or female with a history of COVID with diagnosis confirmed by PCR test.
2. Has been seen at UTMB Post COVID clinic.
3. Minimum of 6 months since diagnosis of COVID by PCR test.
4. Ages 18 to 80 years.
5. Score of 3 or higher on any question 1-3 of the Brief Fatigue Inventory (BFI) questionnaire.
6. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Current COVID infection.
2. Unable to walk unassisted.
3. Significant heart, liver, kidney, blood or respiratory disease.
4. Uncontrolled diabetes mellitus.
5. Any history of a recently (12 months) diagnosed cancer other than a skin cancer (excluding melanoma).
6. Current alcohol or drug abuse.
7. History of psychosis.
8. Pregnancy or become pregnant during the trial.
9. Subjects who are being managed with narcotics will be excluded as the effects of central nervous system depressants may interfere with study test results.
10. Other medical condition or medication administration deemed exclusionary by the study investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Subjects recovered from COVID without lingering symptoms (nPASC)
  2. Subjects with post-COVID syndrome (PASC)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Urban, MD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright TJ, Pyles RB, Sheffield-Moore M, Deer RR, Randolph KM, McGovern KA, Danesi CP, Gilkison CR, Ward WW, Vargas JA, Armstrong PA, Lindsay SE, Zaidan MF, Seashore J, Wexler TL, Masel BE, Urban RJ. Low growth hormone secretion associated with post-acute sequelae SARS-CoV-2 infection (PASC) neurologic symptoms: A case-control pilot study. Mol Cell Endocrinol. 2024 Jan 1;579:112071. doi: 10.1016/j.mce.2023.112071. Epub 2023 Oct 8. PMID 37816478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from May 2021 to May 2022. Subjects for PASC group were recruited from the UTMB post-COVID clinic. Subjects for the nPASC group were recruited from the community. All subjects were required to have a confirmed PCR diagnosis of SARS-CoV-2 at least 6 months prior to enrollment as well as confirmed negative at enrollment. Confirmed SARS-CoV-2 infection dates for subjects ranged from June 2020 to August 2021, before the emergence and dominance of the Omicron variant.
Groups:
- Symptomatic Post-COVID (PASC): Patients with post-acute sequelae of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (PASC)
- Non-symptomatic Post-COVID (nPASC): Patients with that recovered without lingering symptoms after being infected with post-acute sequelae of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
Period: Overall Study
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Started | 10 | 13
Completed | 9 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Symptomatic Post-COVID: 10 patients with Post-COVID syndrome
- Non-symptomatic Post-COVID: 13 patients with that recovered without lingering symptoms after being infected with COVID
- Total: Total of all reporting groups
Arm/Group | Symptomatic Post-COVID | Non-symptomatic Post-COVID | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (9.9) | 46.8 (14.9) | 47.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 12 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Days post-diagnosis [Mean (Standard Deviation); unit: days] | 293.9 (97.1) | 473.0 (145.8) | 395.1 (153.9)
COVID Hospitalization [Count of Participants; unit: Participants] | 2 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] | 164.2 (9.8) | 170.7 (8.8) | 167.9 (9.6)
Weight [Mean (Standard Deviation); unit: kg] | 85.2 (23.0) | 90.3 (16.4) | 88 (19.2)
BMI [Mean (Standard Deviation); unit: (kg/m^2)] | 31.2 (5.9) | 30.9 (4.5) | 31.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Insulin-Like Growth Factor-1 (IGF1)
Description: Insulin-Like Growth Factor-1 (IGF1) will be measured in serum. Results will be reported in ng/mL.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Symptomatic Post-COVID: Patients with Post-COVID syndrome
Arm/Group | Symptomatic Post-COVID | Non-symptomatic Post-COVID
Number analyzed (Participants) | 10 | 13
ng/ml | 142.8 (41.6) | 137.6 (56.7)

2. Primary Outcome: Follicle Stimulating Hormone (FSH)
Description: Follicle Stimulation Hormone (FSH) will be measured in serum.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Symptomatic Post-COVID | Non-symptomatic Post-COVID
Number analyzed (Participants) | 10 | 13
mIU/ml | 38.2 (35.3) | 24.1 (32.7)

3. Primary Outcome: Sex Hormone Binding Globulin (SHBG)
Description: Sex Hormone Binding Globulin (SHBG) will be measured in serum. Results will be reported in nmol/L.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Symptomatic Post-COVID | Non-symptomatic Post-COVID
Number analyzed (Participants) | 10 | 13
nmol/L | 46.4 (25.0) | 97.7 (85.8)

4. Primary Outcome: Total Testosterone
Description: Total testosterone will be measured in serum of male subjects. Results will be reported in ng/dL.
Time Frame: baseline
Population: Testosterone reported in male subjects only
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Symptomatic Post-COVID | Non-symptomatic Post-COVID
Number analyzed (Participants) | 2 | 4
ng/dl | 508.0 (81.2) | 292.5 (53.0)

5. Primary Outcome: Free Testosterone
Description: Free testosterone will be measured in serum of male subjects. Results will be reported in pg/mL.
Time Frame: baseline
Population: Free testosterone measured in males only
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 2 | 4
pg/ml | 27.9 (37.0) | 76.0 (4.6)

6. Primary Outcome: Prolactin
Description: Prolactin will be measured in serum. Results will be reported in ng/mL.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 13
ng/ml | 11.5 (9.5) | 9.5 (4.0)

7. Primary Outcome: Thyroid Stimulating Hormone (TSH)
Description: Thyroid Stimulating Hormone (TSH) will be measured in serum. Results will be reported in mUI/L.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mUI/L
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 13
mUI/L | 2.38 (1.27) | 1.60 (0.95)

8. Primary Outcome: C Reactive Protein (CRP)
Description: C Reactive Protein (CRP) will be measured in serum.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 13
mg/dl | 0.47 (0.46) | 0.38 (0.57)

9. Primary Outcome: Vitamin B12
Description: Vitamin B12 will be measured in serum.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 13
pg/ml | 553.7 (156.4) | 446.1 (254.3)

10. Primary Outcome: Vitamin D 25OH
Description: Vitamin D 25OH will be measured in serum.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 13
ng/ml | 30.6 (8.6) | 41.1 (10.7)

11. Primary Outcome: Glucose Tolerance as Measured by the Oral Glucose Tolerance Test (OGTT) Before Glucose Consumption
Description: Glucose will be measured in serum before (0 minutes) oral consumption of 75g glucose. OGTT will be performed on PASC subjects only.
Time Frame: Before glucose consumption
Population: PASC subjects only
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 0
mg/dl | 91.9 (6.9) |

12. Primary Outcome: Glucose Tolerance as Measured by the Oral Glucose Tolerance Test (OGTT) 120 Minutes After Glucose Consumption
Description: Glucose will be measured in serum at 120 minutes after oral consumption of 75g glucose. OGTT will be performed on PASC subjects only.
Time Frame: 120 minutes after glucose consumption
Population: OGTT will be performed on PASC subjects only.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 0
mg/dl | 150.3 (33.7) |

13. Primary Outcome: Insulin as Measured by the Oral Glucose Tolerance Test (OGTT) Before Glucose Consumption
Description: Insulin will be measured in serum before (0 min) oral consumption of 75g glucose. OGTT will be performed on PASC subjects only.
Time Frame: Before glucose consumption
Population: OGTT will be performed on PASC subjects only. 2 subjects from PASC are missing this analysis.
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 8 | 0
uIU/ml | 7.4 (4.4) |

14. Primary Outcome: Insulin as Measured by the Oral Glucose Tolerance Test (OGTT) 120 Minutes After Glucose Consumption
Description: Insulin will be measured in serum at 120 minutes after oral consumption of 75g glucose. OGTT will be performed on PASC subjects only.
Time Frame: 120 minutes after glucose consumption
Population: OGTT will be performed on PASC subjects only. 2 subjects from the PASC group are missing from analysis for this measure.
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 8 | 0
uIU/ml | 82.0 (46.7) |

15. Primary Outcome: Glucose Derived CO2 as Measured by Breath During the Oral Glucose Tolerance Test (OGTT) 120 Minutes After Glucose Consumption
Description: Glucose derived CO2 will be measured in breath samples at 120 minutes after oral consumption of 75g glucose isotopically labeled with 150 mg [U-13C6] glucose.
  Glucose-derived breath CO2 data are analyzed by measuring the ratios of 13CO2 to 12CO2 in single breath samples using an UBiT-IR300 infrared spectrophotometer (Otsuka Electronics, Hirakata, Osaka, Japan). The UBIT-IR300 calculates the difference in 13CO2 abundance from the baseline breath sample to each timed sample and expresses this as per mille delta over baseline (%DOB).
  OGTT will be performed on PASC subjects only.
Time Frame: 120 minutes after glucose consumption
Population: OGTT will be performed on PASC subjects only.
Measure: Mean (Standard Deviation); unit: %DOB
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 0
%DOB | 40.9 (12.6) |

16. Primary Outcome: Sleep Quality as Measured by Pittsburgh Sleep Quality Index
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality.
Time Frame: baseline
Population: 1 PASC subject missing from analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
score on a scale | 11.1 (4.0) | 4.5 (2.8)

17. Primary Outcome: Growth Hormone as Measured by Glucagon Stimulation Test Before Glucagon Administration
Description: Growth hormone secretion will be measured using the glucagon stimulation test. Serum will be collected for the baseline (time: 0 minutes) to test for levels of human growth hormone. 1 mg glucagon (for subjects over 90 kg, 1.5 mg glucagon) will be injected intramuscularly (IM) in the deltoid muscle of the subject and blood will be drawn at specified time points.
  Results will be reported as ng/mL.
Time Frame: Before glucagon administration
Population: One PASC patient is missing from this measure
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
ng/ml | 0.4 (0.6) | 0.9 (0.8)

18. Primary Outcome: Growth Hormone as Measured by Glucagon Stimulation Test 90 Minutes After Glucagon Administration
Description: Growth hormone secretion will be measured using the glucagon stimulation test. Serum will be collected at time point 90 minutes after glucagon injection to test for levels of human growth hormone.
  Results will be reported as ng/mL.
Time Frame: 90 minutes after glucagon administration
Population: One PASC patient is missing from this measure
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
ng/ml | 0.6 (0.5) | 1.6 (3.5)

19. Primary Outcome: Growth Hormone as Measured by Glucagon Stimulation Test 120 Minutes After Glucagon Administration
Description: Growth hormone secretion will be measured using the glucagon stimulation test. Serum will be collected at timepoint 120 minutes after glucagon injection to test for levels of growth hormone.
  Results will be reported as ng/mL.
Time Frame: 120 minutes after glucagon administration
Population: One PASC patient is missing from this measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
ng/ml | 2.2 (2.5) | 5.6 (6.0)

20. Primary Outcome: Growth Hormone as Measured by Glucagon Stimulation Test 150 Minutes After Glucagon Administration
Description: Growth hormone secretion will be measured using the glucagon stimulation test. Serum will be collected at timepoint 150 minutes after glucagon injection to test for levels of growth hormone.
  Results will be reported as ng/mL.
Time Frame: 150 minutes after glucagon administration
Population: One PASC patient is missing from this measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
ng/ml | 2.6 (2.1) | 5.8 (3.5)

21. Primary Outcome: Growth Hormone as Measured by Glucagon Stimulation Test 180 Minutes After Glucagon Administration
Description: Growth hormone secretion will be measured using the glucagon stimulation test. Serum will be collected at timepoint 180 minutes after glucagon injection to test for levels of growth hormone.
  Results will be reported as ng/mL.
Time Frame: 180 minutes after glucagon administration
Population: One PASC patient is missing from this measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
ng/ml | 2.3 (1.9) | 3.0 (2.1)

22. Primary Outcome: Basal Metabolic Rate as Measured by Resting Energy Expenditure
Description: Resting Energy Expenditure will be measured by capturing the expired breath of subjects while at rest with a metabolic cart over a 30 minute time period. Data from the first 5 minutes will be discarded and the remaining 25 minutes of data will be averaged to calculate the resting energy expenditure. Data will be reported as kilocalories/day
  Procedure will be performed on PASC subjects only.
Time Frame: baseline
Population: PASC patients only. 2 patients from the PASC group are missing from measure.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 8 | 0
kcal/day | 1489.2 (257.7) |

23. Primary Outcome: Cortisol as Measured by the Adrenocorticotropic Hormone Stimulation Test (ACTH) Before Cortrosyn Administration
Description: Cortisol secretion will be measured using the ACTH stimulation test. Serum will be collected for the baseline (time: 0 minutes) to test for levels of cortisol. 0.25 mg Cortrosyn will be administered and additional serum (3.5 mL) will be collected at specified time points.
  Results will be reported as ug/dL. Procedure will be performed on PASC subjects only.
Time Frame: Before Cortrosyn administration
Population: PASC patients only.
  1 PASC patient is missing from measure.
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 0
ug/dl | 5.3 (2.3) |

24. Primary Outcome: Cortisol as Measured by the Adrenocorticotropic Hormone Stimulation Test (ACTH) 30 Minutes After Cortrosyn Administration
Description: Cortisol secretion will be measured using the ACTH stimulation test. Serum will be collected at time point 30 minutes after Cortrosyn administration to test for levels of cortisol. Procedure will be performed on PASC subjects only.
  Results will be reported as ug/dL.
Time Frame: 30 minutes after Cortrosyn administration
Population: PASC patients only
  1 PASC patient missing from measure
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 0
ug/dl | 17.9 (2.4) |

25. Primary Outcome: Cortisol as Measured by the Adrenocorticotropic Hormone Stimulation Test (ACTH) 60 Minutes After Cortrosyn Administration
Description: Cortisol secretion will be measured using the ACTH stimulation test. Serum will be collected at time point 60 minutes after Cortrosyn administration to test for levels of cortisol.
  Results will be reported as ug/dL. Procedure will be performed on PASC subjects only.
Time Frame: 60 minutes after Cortrosyn administration
Population: PASC patients only.
  1 PASC patient missing from measure.
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 0
ug/dl | 21.7 (2.6) |

26. Primary Outcome: Cognitive Function as Measured by Montreal Cognitive Assessment
Description: The Montreal Cognitive Assessment (MoCA) will be used to assess cognition.
  The Montreal Cognitive Assessment (MoCA) is a rapid assessment of cognition. The MoCA consists of 9 questions with the following subcategories: visuospatial/executive, naming, memory, language, abstraction, delayed recall and orientation. The MoCA has been used extensively to detect cognitive impairment in many conditions, including head trauma. Version 7.1 will be used. Scores range from 0 to 30, higher score being a better outcome.
Time Frame: baseline
Population: 1 PASC patient missing from measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
units on a scale | 27.0 (2.5) | 27.9 (2.8)

27. Primary Outcome: Gastrointestinal Health Measured by the Gastrointestinal Symptom Rating Scale
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort). The average of the scores for all 15 items is regarded as the GSRS total score. A higher score indicates a worse outcome.
Time Frame: baseline
Population: 1 PASC patient is missing from this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
units on a scale | 2.5 (1.0) | 1.4 (0.4)

28. Primary Outcome: Fatigue as Measured by the Multidimensional Fatigue Symptom Inventory
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: baseline
Population: 1 PASC patient is missing from this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
units on a scale | 31.0 (17.3) | -14.0 (7.4)

29. Primary Outcome: Symptoms of Growth Hormone Deficiency Measured by the Questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults
Description: Symptoms of growth hormone deficiency will be measured using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms.
Time Frame: baseline
Population: 1 PASC patient is missing from this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
units on a scale | 13.6 (7.0) | 2.4 (5.1)

30. Primary Outcome: Depression Measured by the Beck Depression Inventory-II
Description: The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Time Frame: baseline
Population: 1 PASC patient is missing from this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 9 | 13
units on a scale | 16.8 (10.7) | 2.2 (5.4)

31. Secondary Outcome: Free T4
Description: Free T4 measured at baseline
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
Number analyzed (Participants) | 10 | 13
ng/dl | 1.05 (0.16) | 1.19 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, an average of 3 weeks.
Arm/Group | Symptomatic Post-COVID (PASC) | Non-symptomatic Post-COVID (nPASC)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04860869/Prot_SAP_000.pdf